CLINICAL TRIAL: NCT04449536
Title: Cysteine-lowering Treatment With Mesna Against Obesity: Phase I Dose-finding Study
Brief Title: Cysteine-lowering Treatment With Mesna
Acronym: CYLOB
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Oslo (Other)
Collaborators: Oslo University Hospital (Other); University of Oxford (Other)
Responsible Party: Principal Investigator, Kathrine Vinknes, Researcher and Project manager, University of Oslo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EudraCT: 2019-003412-32
Record Dates: First submitted 2020-06-15; First posted 2020-06-29 (Actual); Last update posted 2022-05-19 (Actual); Status verified 2022-05

CONDITIONS: Obesity; Drug Effect
Keywords: Cysteine; Phase 1; Mesna
MeSH Terms: conditions — Obesity | interventions — Mesna

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mesna (Experimental): Administration of a single oral dose of 400 mg, 800 mg, 1200 mg or 1600 mg
  Interventions: Drug: Mesna

INTERVENTIONS:
Drug: Mesna — Administration of a single oral dose, using film-coated tablets of either 400 mg or 600 mg or a combination of maximum 3 tablets up to a maximum of 1600 mg
  Other Names: Uromitexan

SUMMARY:
The primary objective of this study is to determine the efficacy of the drug Mesna® (Uromitexan) in healthy participants with overweight or obesity with respect to change in plasma concentrations of total cysteine, following single ascending doses of oral Mesna.

DETAILED DESCRIPTION:
In both animal experiments and human studies, cysteine in the blood is strongly associated with obesity. In rodents, changes in cysteine induced by dietary means are accompanied by changes in fat mass.

In this phase I, single ascending dose study the investigators will determine the effects of Mesna in healthy volunteers with overweight and obesity with focus on its effects on plasma total cysteine concentrations. The aim of this dose-finding clinical trial is to determine the lowest single oral Mesna dose that will lower plasma total cysteine concentrations by 30% using pharmacokinetic (PK)/ pharmacodynamic (PD) modelling. The investigators will further evaluate the effect of Mesna on plasma cysteine fractions and related metabolites, urinary cysteine excretion, safety and adverse drug reactions, and plasma biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* BMI between BMI 27-40 kg/m2
* Age between 18-55 years
* Male
* Healthy as determined by medical evaluation, medical history, physical examination, 12-lead ECG, and laboratory tests

Exclusion Criteria:

* Presence of chronic disease
* Chronic drug use
* Past or intended use of over-the-counter or prescription medication including herbal medications within 14 days prior to dosing
* Veganism
* Strenuous physical activity ≥3 times every week
* Smoking

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2020-11-02 (Actual); Primary Completion 2021-10-21 (Actual); Study Completion 2021-10-21 (Actual)

PRIMARY OUTCOMES:
Change in plasma total cysteine concentrations following single ascending doses of oral Mesna. | Several intervals during the first 12 hours after Mensa administration, and a fasting sample on days 2 and 3
  Nadir plasma total cysteine concentrations

SECONDARY OUTCOMES:
Pharmacokinetic parameter - maximum plasma concentration (Cmax) | Several intervals during the first 12 hours after Mesna administration, and a fasting sample on days 2 and 3
  Maximum plasma Mesna concentration (Cmax) after a single oral Mesna dose
Pharmacokinetic parameter - time to maximum plasma concentration (Tmax) | Several intervals during the first 12 hours after Mesna administration, and a fasting sample on days 2 and 3
  Time to maximum plasma Mesna concentration (Tmax) after a single oral Mesna dose
Pharmacokinetic parameter - area under the plasma concentration-time curve (AUC) | Several intervals during the first 12 hours after Mesna administration, and a fasting sample on days 2 and 3
  Area under the plasma Mesna concentration-time curve (AUC)0-inf after a single oral Mesna dose
Pharmacokinetic parameter - elimination rate constant (Kel) | Several intervals during the first 12 hours after Mesna administration, and a fasting sample on days 2 and 3
  Elimination rate constant (Kel) for Mesna after a single oral Mesna dose
Pharmacokinetic parameter - dose linearity | Several intervals during the first 12 hours after Mesna administration, and a fasting sample on days 2 and 3
  Dose linearity of Mesna after a single oral Mesna dose
Change in plasma cystine, free reduced cysteine, and protein bound cysteine | Several intervals during the first 12 hours after Mesna administration, and a fasting sample on days 2 and 3
  Estimated AUCs
Urine excretion of cysteine | During the first 24 hours after Mesna administration
  Cumulative and fractional excretion of total cysteine and Mesna
Safety of Mesna | During the first 5 days after Mesna administration
  Occurrence/prevalence of side effects, adverse events, and serious adverse events

OTHER OUTCOMES:
Changes in plasma and urine sulfur amino acids and related metabolites | Several intervals during the first 12 hours after Mesna administration, and a fasting sample on days 2 and 3
  Estimated AUCs
Changes in plasma biomarker concentration - glucose | During the first 24 hours after Mesna administration, and a fasting sample on days 2 and 3
  Estimated AUC
Changes in plasma biomarker concentration - insulin | During the first 24 hours after Mesna administration, and a fasting sample on days 2 and 3
  Estimated AUC
Changes in plasma biomarker concentration - lipids | During the first 24 hours after Mesna administration, and a fasting sample on days 2 and 3
  Estimated AUC

CONTACTS AND LOCATIONS:
Overall Officials: Kjetil Retterstøl, MD, PhD, Principal Investigator — University of Oslo
Locations (1):
- University of Oslo, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No
Data that support the findings of this study may be available upon reasonable request from qualified users.